CLINICAL TRIAL: NCT00625885
Title: Multicenter ACL Revision Study (MARS)
Acronym: MARS
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kurt P. Spindler, Adjoint Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 070110; R01AR060846 (NIH)
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: Anterior Cruciate Ligament/injuries; Anterior Cruciate Ligament/surgery; Knee injuries/surgery; Outcomes research; Prospective Studies
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the effects of modifiable risk factors on patient-reported quality of life, physical activity levels, and risk of early osteoarthritis following revision anterior cruciate ligament (ACL) reconstruction.

The investigators hypothesize that modifiable variables exist at the time of revision ACL reconstruction (e.g., cause of failure, current graft source and type, surgical exposure, and femoral and tibial tunnel position) which will be predictors of patient-reported outcomes.

DETAILED DESCRIPTION:
Injury to the anterior cruciate ligament (ACL) results in a threat to an active lifestyle and exposes the patient to risk of osteoarthritis. ACL reconstruction is typically chosen by individuals to allow a return to their previous work and sports activities. The results of primary ACL reconstruction have in general been good at restoring functional stability. Primary ACL reconstruction has a graft failure rate ranging from approximately 2%-8%. Consensus amongst surgeons and low-level evidence (retrospective case series) indicate a worse outcome following revision ACL reconstruction compared to primary reconstruction. The typical surgeon performs less than 10 revision ACL reconstructions per year. Thus, the ability of any single surgeon or small group of surgeons to accumulate enough cases to effectively analyze predictors for worse outcome is impossible.

With this in mind, the Multi-Center ACL Revision Study (MARS) group was established as a multi-center surgeon group to perform a prospective longitudinal cohort analysis of revision ACL reconstruction. This is a mixed group of academic and private practice physicians and has been supported and endorsed by the American Orthopedic Society for Sports Medicine (AOSSM).

This study focuses on the predictors for ACL revision outcome at 2, 6,10 and 20 years following a patient's revision ACL reconstruction. This will be accomplished by three Specific Aims. Specific Aim 1 will determine the independent predictors of patient-reported quality of life, utilizing a general (SF-36) and knee-specific (Knee Injury and Osteoarthritis Outcome Score - KOOS) validated outcome instrument. Specific Aim 2 will determine the independent predictors of sports function utilizing three validated outcome instruments (the Marx activity level, International Knee Documentation Committee Subjective form - IKDC, and the KOOS sports and recreation subscale). Specific Aim 3 will identify those independent modifiable predictors measured at the time of the revision ACL reconstruction associated with symptoms of knee osteoarthritis at up to 20 years post-surgery. Symptoms will be quantified using the validated survey instrument the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Once the predictors for these worse outcomes are identified, surgeons can be educated in potential modifiable variables to improve the outcome.

ELIGIBILITY:
Inclusion Criteria:

* All ACL-deficient candidates presenting to the clinic, between the ages of 12† and 65, scheduled to have a revision ACL reconstruction by a participating (MARS Study) surgeon.
* All participants must have undergone a primary ACL reconstruction in the past and are currently identified as having experienced failure of their primary ACL reconstruction, as defined by either MRI, knee laxity (KT > 5mm), a positive pivot shift or Lachman's, functional instability, and/or by arthroscopic confirmation.
* All ACL-deficient patients seeking a revision ACL reconstruction that have either partial (Grade I or II) and/or complete (Grade III) simultaneous ligamentous injuries to the collateral ligaments (MCL or LCL) and/or the posterior cruciate ligament (PCL) will also be included.
* Non-operative treatment of patients with ACLR failure are also eligible to participate.
* The following graft types will be the only ones accepted for inclusion:

  * any autograft
  * Fresh-frozen allografts from a single donor source (Musculoskeletal Transplant Foundation (MTF); Edison, NJ). These grafts should consist of either:

    * bone-patellar tendon-bone
    * tibialis anterior/posterior
    * achilles tendon

Exclusion Criteria:

* Patients presenting with prior infection, arthrofibrosis, or regional pain syndrome.
* Subjects will be excluded if their allograft source does not come from MTF.
* Patients unwilling or unable to complete their repeat questionnaire two years after their initial visit.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All ACL-deficient candidates scheduled for a revision ACL reconstruction at one of the participating MARS sites.
Sampling Method: Non-Probability Sample
Enrollment: 1234 (Actual)
Dates: Start 2006-03-26 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Graft re-rupture | 2, 6, 10, and 20 years after revision ACL surgery

SECONDARY OUTCOMES:
Patient based outcome measures | 2, 6,10, and 20 years after revision ACL surgery
  Activity level (as measured by the Marx activity scale). Sports function (as measured by the KOOS and IKDC). Pain and swelling (as measured by the WOMAC).

CONTACTS AND LOCATIONS:
Overall Officials: Rick W. Wright, M.D., Principal Investigator — Vanderbilt University Medical Center; Kurt P. Spindler, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (49):
- United States (47):
  - Scripps Memorial Hospital (OrthoCal Healthcare), La Jolla, California
  - University of California - Los Angeles (UCLA), Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Orthopaedic Associates of Aspen and Glenwood, Aspen, Colorado
  - University of Colorado, Boulder, Colorado
  - Connecticut Children's Medical Center, Farmington, Connecticut
  - University of Connecticut Health Center, Farmington, Connecticut
  - UHZ Sports Medicine Institute, Coral Gables, Florida
  - Intermountain Orthopaedics, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Methodist Sports Medicine Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Cheaspeake Orthopaedics and Sports Medicine Center, Glen Burnie, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Regions Hospital (Health Partners Research Foundation), Saint Paul, Minnesota
  - Washington University at St. Louis, St Louis, Missouri
  - Bridger Orthopaedic and Sports Medicine, Bozeman, Montana
  - New Hamphsire Knee Center, Holderness, New Hampshire
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Princeton Orthopaedic Associates, Princeton, New Jersey
  - University of Buffalo, Buffalo, New York
  - NYU School of Medicine, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Manhattan Orthopaedics, P.C., New York, New York
  - Keller Army Community Hospital - USMA, West Point, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Perry Orthopaedics and Sports Med (Carolinas Healthcare System), Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Slocum Research and Education Foundation, Eugene, Oregon
  - Orthopaedic and Fracture Clinic, Portland, Oregon
  - The Rothman Institute / Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Booth, Bartolozzi, Balderston Orthopaedics, Philadelphia, Pennsylvania
  - Orthopaedic Institute, Sioux Falls, South Dakota
  - Southeastern Orthopaedics / Knoxville Orthopaedic Clinic, Knoxville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - W.B. Carroll Memorial Clinic, Dallas, Texas
  - San Antonio Orthopaedic Group, San Antonio, Texas
  - University of Vermont College of Medicine, Burlington, Vermont
  - National Sports Medicine Institute, Lansdowne, Virginia
  - Town Center Orthopaedic Associates, Reston, Virginia
  - Commonwealth Orthopaedics and Rehabilitation, Vienna, Virginia
  - Inland Orthopaedics/Washington State University, Pullman, Washington
- Canada (2):
  - Royal Columbian Hospital (FraserHealth), New Westminster, British Columbia
  - Fowler Kennedy Sports Medicine Clinic/Univ. of Western Ontario, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] MARS Group; Vasavada K, Vasavada V, Moran J, Devana S, Lee C, Hame SL, Jazrawi LM, Sherman OH, Huston LJ, Haas AK, Allen CR, Cooper DE, DeBerardino TM, Spindler KP, Stuart MJ, Ned Amendola A, Annunziata CC, Arciero RA, Bach BR Jr, Baker CL 3rd, Bartolozzi AR, Baumgarten KM, Berg JH, Bernas GA, Brockmeier SF, Brophy RH, Bush-Joseph CA, Butler V JB, Carey JL, Carpenter JE, Cole BJ, Cooper JM, Cox CL, Creighton RA, David TS, Dunn WR, Flanigan DC, Frederick RW, Ganley TJ, Gatt CJ Jr, Gecha SR, Giffin JR, Hannafin JA, Lindsay Harris N Jr, Hechtman KS, Hershman EB, Hoellrich RG, Johnson DC, Johnson TS, Jones MH, Kaeding CC, Kamath GV, Klootwyk TE, Levy BA, Ma CB, Maiers GP 2nd, Marx RG, Matava MJ, Mathien GM, McAllister DR, McCarty EC, McCormack RG, Miller BS, Nissen CW, O'Neill DF, Owens BD, Parker RD, Purnell ML, Ramappa AJ, Rauh MA, Rettig AC, Sekiya JK, Shea KG, Slauterbeck JR, Smith MV, Spang JT, Svoboda SJ, Taft TN, Tenuta JJ, Tingstad EM, Vidal AF, Viskontas DG, White RA, Williams JS Jr, Wolcott ML, Wolf BR, Wright RW, York JJ. A Novel Machine Learning Model to Predict Revision ACL Reconstruction Failure in the MARS Cohort. Orthop J Sports Med. 2024 Nov 14;12(11):23259671241291920. doi: 10.1177/23259671241291920. eCollection 2024 Nov. PMID 39555321
- [Derived] MARS Group; Cooper DE, Dunn WR, Huston LJ, Haas AK, Spindler KP, Allen CR, Anderson AF, DeBerardino TM, Lantz BBA, Mann B, Stuart MJ, Albright JP, Amendola AN, Andrish JT, Annunziata CC, Arciero RA, Bach BR Jr, Baker CL 3rd, Bartolozzi AR, Baumgarten KM, Bechler JR, Berg JH, Bernas GA, Brockmeier SF, Brophy RH, Bush-Joseph CA, Butler V JB, Campbell JD, Carey JL, Carpenter JE, Cole BJ, Cooper JM, Cox CL, Creighton RA, Dahm DL, David TS, Flanigan DC, Frederick RW, Ganley TJ, Garofoli EA, Gatt CJ Jr, Gecha SR, Giffin JR, Hame SL, Hannafin JA, Harner CD, Harris NL Jr, Hechtman KS, Hershman EB, Hoellrich RG, Hosea TM, Johnson DC, Johnson TS, Jones MH, Kaeding CC, Kamath GV, Klootwyk TE, Levy BA, Ma CB, Maiers GP 2nd, Marx RG, Matava MJ, Mathien GM, McAllister DR, McCarty EC, McCormack RG, Miller BS, Nissen CW, O'Neill DF, Owens BD, Parker RD, Purnell ML, Ramappa AJ, Rauh MA, Rettig AC, Sekiya JK, Shea KG, Sherman OH, Slauterbeck JR, Smith MV, Spang JT, Svoboda SJ, Taft TN, Tenuta JJ, Tingstad EM, Vidal AF, Viskontas DG, White RA, Williams JS Jr, Wolcott ML, Wolf BR, York JJ, Wright RW. Physiologic Preoperative Knee Hyperextension Is a Predictor of Failure in an Anterior Cruciate Ligament Revision Cohort: A Report From the MARS Group. Am J Sports Med. 2018 Oct;46(12):2836-2841. doi: 10.1177/0363546518777732. Epub 2018 Jun 8. PMID 29882693
- [Derived] MARS Group. Meniscal and Articular Cartilage Predictors of Clinical Outcome After Revision Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2016 Jul;44(7):1671-9. doi: 10.1177/0363546516644218. Epub 2016 May 9. PMID 27161867